CLINICAL TRIAL: NCT02587195
Title: A National, Multi-center Study to Evaluate the Safety of Long Term Treatment With Teriflunomide 14 mg Once Daily in Patients With a First Clinical Episode Suggestive of Multiple Sclerosis in a Long-term Extension Period
Brief Title: A Study to Evaluate the Safety of Long Term Treatment With Teriflunomide 14 mg Once Daily in Patients With a First Clinical Episode Suggestive of Multiple Sclerosis in a Long-term Extension Period
Acronym: TERICIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-PP-06
Record Dates: First submitted 2015-09-22; First posted 2015-10-27 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Teriflunomide (Experimental): Teriflunomide 14 mg Once Daily
  Interventions: Drug: Teriflunomide

INTERVENTIONS:
Drug: Teriflunomide

SUMMARY:
National, multicenter study:

The study consists of 3 periods:

1. A baseline visit to confirm that patient is still in CIS status. All patients will be clinically evaluated for CDMS and an MRI (less than 2 months) will be analyzed to exclude MS patients according to 2010 Mc Donald's criteria.
2. Treatment period with timed evaluations
3. Post-treatment period: 4 weeks, with 2 visits following study drug discontinuation and accelerated elimination procedure. All patients who discontinue the study drug and according to investgator's decision, will perform the accelerated elimination procedure and the post- accelerated elimination visits (at 2 and 4 weeks after the end of treatment (EOT).

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in TOPIC study and extension of TOPIC study and currently treated in French extension of TOPIC study who did not convert into MS.
* A baseline MRI scan (performed less than 2 months before baseline Visit ) confirming that patient is still in CIS status.

Exclusion Criteria:

* Contraindication for MRI,
* Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major systemic disease or procedure/medication making implementation of the protocol or interpretation of the study results difficult or that would put the patient at risk by participating in the study
* Patients with a congenital or acquired severe immunodeficiency, a history of cancer (except for basal or squamous cell skin lesions which have been surgically excised, with no evidence of metastasis), lymphoproliferative disease, or any patient who has received lymphoid irradiation
* Known history of active tuberculosis not adequately treated
* Persistent significant or severe infection
* History of drug or alcohol abuse
* Patients must not have used Adrenocorticotrophic hormone (ACTH) or systemic corticosteroids for 2 weeks prior to inclusion
* Prior use within 4 weeks before inclusion or concomitant use of cholestyramine
* Prior or concomitant use of cladribine, mitoxantrone, or other immunosuppressant agents such as azathioprine, cyclophosphamide, cyclosporin, methotrexate or mycophenolate
* Prior or concomitant use of interferons, cytokine therapy, glatiramer acetate or intravenous immunoglobulins
* Prior or concomitant use of natalizumab (Tysabri®)
* Pregnant or breast-feeding women
* Women of childbearing potential not protected by effective contraceptive method of birth control and/or who are unwilling or unable to be tested for pregnancy.
* Women wishing to become pregnant during the course of the trial
* Patients with significantly impaired bone marrow function or significant anemia, leukopenia, or thrombocytopenia
* Human immunodeficiency virus (HIV) positive patient
* Persisting elevations (confirmed by retest) of serum amylase or lipase greater than 2-fold the upper limit of normal
* Known history of chronic pancreatic disease or pancreatitis
* Liver function impairment or persisting elevations (confirmed by retest) of serum glutamic pyruvic transaminase (SGPT/ALT), serum glutamic oxaloacetic transaminase (SGOT/AST), or direct bilirubin greater than 1.5-fold the upper limit of normal
* Known history of active hepatitis
* Hypoproteinemia (e.g., in case of severe liver disease or nephrotic syndrome) with serum albumin < 3.0 g/dL
* Moderate to severe impairment of renal function, as shown by serum creatinine > 133 μmol/L (or > 1.5 mg/dL)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse event reporting | throughout study completion an average of 6 months
  evaluation of safety and tolerability of teriflunomide 14mg per day
Adverse Events That Are Related to Treatment | throughout study completion an average of 6 months

SECONDARY OUTCOMES:
Conversion based on MRI | throughout study completion an average of 6 months
  Conversion to definite MS based on MRI data as defined by the demonstration of dissemination of MRI lesions in time (based on the 2010 revised McDonald criteria) within 3 years
Conversion based on Clinical evaluation | throughout study completion an average of 6 months
  Conversion to clinically definite MS based on clinical evaluation and annualized relapse rate (ARR), defined as number of relapses per patient-year
Conversion based on annualized relapse rate (ARR) | throughout study completion an average of 6 months
  Conversion to clinically definite MS based on clinical evaluation and annualized relapse rate (ARR), defined as number of relapses per patient-year
volume of abnormal brain tissue on MRI | 3 years
Disability progression defined as a 1.0-point increase in EDSS score | confirmed after at least 12 weeks
  to disability progression (12 weeks), defined as a 1.0-point increase in EDSS score (or 0.5-point increase for baseline EDSS >5.5) confirmed after at least 12 weeks
Proportion of disability-free subjects as assessed by the EDSS | throughout study completion an average of 1 year
  Proportion of disability-free subjects as assessed by the EDSS
Fatigue Impact Scale | throughout study completion an average of 1 year
  Patient-reported fatigue based on the Fatigue Impact Scale
Quality of life using SF-36 | throughout study completion an average of 1 year

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU de Besançon, Besançon
  - CHU de Lille, Lille
  - CHU de Montpellier, Montpellier
  - CHU de Nice, Nice
  - CHU de Strasbourg, Strasbourg